CLINICAL TRIAL: NCT00007150
Title: Studies of Phlebotomy Therapy in Hereditary Hemochromatosis
Brief Title: Treatment of Hemochromatosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 010045; 01-CC-0045
Record Dates: First submitted 2000-12-09; First posted 2000-12-11 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-06

CONDITIONS: Hemochromatosis
Keywords: Phlebotomy Therapy; Hemochromatosis; Iron Overload; Hereditary Hemochromatosis; Blood Donation
MeSH Terms: conditions — Hemochromatosis; Iron Overload | interventions — Phlebotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/HH patients (Other): HH patients
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Therapeutic phlebotomy, the periodic, frequent removal of the iron contained in the hemoglobin of red blood cells.

SUMMARY:
This study will evaluate the effectiveness of a test called MCV in guiding phlebotomy (blood drawing) therapy in patients with hemochromatosis an inherited disorder that causes too much iron to be absorbed by the intestine. The excess damages body tissues, most severely in the liver, heart, pancreas and joints. Because iron is carried in the hemoglobin of red blood cells, removing blood can effectively lower the body s iron stores.

Patients with hemochromatosis undergo weekly phlebotomy treatments (1 pint per session) to deplete iron stores. This usually requires 10 to 50 treatments, after which blood is drawn every 8 to 12 weeks to prevent a re-build up of iron. A test that measures ferritin a protein involved in storing iron is commonly used to guide phlebotomy therapy in hemochromatosis patients. This study will compare the usefulness of the ferritin test with that of MCV, which measures red blood cell size, in guiding phlebotomy therapy. In addition, the study will 1) examine whether keeping iron levels low during maintenance therapy can help heal severe liver disease and improve arthritis in affected patients, and 2) design a system for making blood collected from hemochromatosis donors available for transfusion into other patients.

Patients 15 years and older with diagnosed hemochromatosis or very high iron levels suggesting possible hemochromatosis may be eligible for this study. Candidates will have a history, physical evaluation, review of medical records and blood tests, and complete a symptoms questionnaire. Participants will have the following procedures:

* Phlebotomy therapy every 1 to 2 weeks, depending on iron levels
* Blood sample collection for blood cell counts and iron studies at every phlebotomy session
* Blood sample collection (about 2 tablespoons) every 1 to 2 weeks after iron stores have been depleted
* Phlebotomy every 8 to 12 weeks after iron stores are used up to prevent re-build up of excess iron

With each blood donation that will be made available for transfusion to other patients, participants will answer the same health history screening questions and undergo the same blood tests given to all regular volunteer blood donors. These include screening for the HIV and hepatitis viruses and for syphilis.

Patients who meet height and weight requirements may be asked to consider "double red cell" donations using apheresis. In this procedure, whole blood is collected through a needle placed in an arm vein, similar to routine phlebotomy. The blood then circulates through a machine that separates it into its components. The red cells are removed and the rest of the blood is returned to the body, either through the same needle or through a second needle in the other arm. Patients who have very high iron levels or an enlarged liver will be offered evaluation by the NIH Liver Service. Those judged to be at increased risk for cirrhosis may be advised to undergo a liver biopsy. If cirrhosis is found, the patient will be asked to consider a repeat biopsy after 3 to 5 years of continuous iron depletion to see if scarring has improved. Patients with arthritis will be offered evaluation by the NIH Arthritis Service and, depending on symptoms, may be advised to have X-ray studies or a joint biopsy.

...

DETAILED DESCRIPTION:
Hereditary hemochromatosis (HH) occurs in 1 in every 200-250 individuals of northern European descent, and is the most common inherited disease in this population. Although the molecular pathophysiology remains incompletely understood, a homozygous mutation in the HFE gene (Cys282Tyr) is observed in nearly 100% of clinically confirmed cases. The clinical manifestations of HH are due to inappropriately increased iron absorption with excessive iron deposition in the liver, heart, endocrine organs, and joints.

Phlebotomy treatment, with removal of iron contained in the hemoglobin of red cells, is the only effective therapy for HH. Phlebotomy therapy relieves many of the symptoms of iron-mediated tissue damage and prevents progression to cirrhosis. However, published laboratory guidelines for monitoring phlebotomy therapy are based on retrospective data, and in general allow a moderate level of iron overload to persist during maintenance therapy. Since 1987, the DTM has piloted the use of the red cell mean corpuscular volume (MCV), in conjunction with the hemoglobin, as a prospective guide to phlebotomy therapy in a small cohort of HH patients. In contrast to other retrospectively-derived guidelines, this simple, inexpensive, physiologic method was found to be a precise indicator of iron-limited erythropoiesis, and could be easily applied to adjust the pace of phlebotomy and prevent excess iron reaccumulation.

Although the majority of persons with HH meet eligibility criteria for allogeneic blood donation, until recently regulatory guidelines restricted the use of therapeutically withdrawn blood for transfusion. New regulations now permit increased flexibility in the use of such units for this purpose. The purposes of this protocol are: (1) to prospectively study the genotypic and phenotypic response to phlebotomy therapy in HH patients using the MCV/hemoglobin monitoring guide, and to validate the use of this guide in a large study cohort; (2) to evaluate the course of severe hepatic disease and rheumatologic symptoms following sustained iron depletion; and (3) to establish the safety and efficacy and document the operational issues inherent in a program to collect therapeutically withdrawn blood for use in allogeneic transfusion. These goals have as their combined target the establishment of the simplest, safest system for donor processing, phlebotomy management, and transfusion of blood drawn from HH subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Confirmed diagnosis of HH, defined by the following HFE genotypes: C282Y/C282 or C282Y/H63D. Up to 50 percent of the total study population may have received prior phlebotomy therapy.

Elevated transferrin saturation and/or ferritin level, but diagnosis of HH not yet confirmed by genotype or liver biopsy.

Elevated transferrin saturation and/or ferritin level without genotype findings listed above, but with elevated hepatic iron index on liver biopsy.

Family member screening (unknown HH phenotype or genotype)

EXCLUSION CRITERIA:

Age less than 15 years.

Pregnancy.

Patients requiring therapeutic phlebotomy for reasons other than iron overload (polycythemia vera).

Patients with iron overload not due to HH (e.g. hepatitis C infection, porphyria cutanea tarda, Wilson s disease, alpha-1-antitrypsin deficiency, alcohol abuse).

Other medical illness or condition which, in the opinion of the Investigators, may contraindicate participation due to risk to patient or to Donor Center.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MCV drops 1-3% below baseline | 4 to 12 months after starting phlebotomy therapy
  Response to phlebotomy therapy in HH patients, as evidenced by iron-depletion

CONTACTS AND LOCATIONS:
Overall Officials: Kamille A West-Mitchell, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lucotte G. Celtic origin of the C282Y mutation of hemochromatosis. Blood Cells Mol Dis. 1998 Dec;24(4):433-8. doi: 10.1006/bcmd.1998.0212. PMID 9851897
- [Background] Feder JN, Tsuchihashi Z, Irrinki A, Lee VK, Mapa FA, Morikang E, Prass CE, Starnes SM, Wolff RK, Parkkila S, Sly WS, Schatzman RC. The hemochromatosis founder mutation in HLA-H disrupts beta2-microglobulin interaction and cell surface expression. J Biol Chem. 1997 May 30;272(22):14025-8. doi: 10.1074/jbc.272.22.14025. PMID 9162021
- [Background] Feder JN, Gnirke A, Thomas W, Tsuchihashi Z, Ruddy DA, Basava A, Dormishian F, Domingo R Jr, Ellis MC, Fullan A, Hinton LM, Jones NL, Kimmel BE, Kronmal GS, Lauer P, Lee VK, Loeb DB, Mapa FA, McClelland E, Meyer NC, Mintier GA, Moeller N, Moore T, Morikang E, Prass CE, Quintana L, Starnes SM, Schatzman RC, Brunke KJ, Drayna DT, Risch NJ, Bacon BR, Wolff RK. A novel MHC class I-like gene is mutated in patients with hereditary haemochromatosis. Nat Genet. 1996 Aug;13(4):399-408. doi: 10.1038/ng0896-399. PMID 8696333
- [Background] Leitman SF, Browning JN, Yau YY, Mason G, Klein HG, Conry-Cantilena C, Bolan CD. Hemochromatosis subjects as allogeneic blood donors: a prospective study. Transfusion. 2003 Nov;43(11):1538-44. doi: 10.1046/j.1537-2995.2003.00570.x. PMID 14617312
- [Derived] Wang X, Mendelsohn L, Rogers H, Leitman S, Raghavachari N, Yang Y, Yau YY, Tallack M, Perkins A, Taylor JG 6th, Noguchi CT, Kato GJ. Heme-bound iron activates placenta growth factor in erythroid cells via erythroid Kruppel-like factor. Blood. 2014 Aug 7;124(6):946-54. doi: 10.1182/blood-2013-11-539718. Epub 2014 Jun 10. PMID 24916507
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-CC-0045.html